CLINICAL TRIAL: NCT02809950
Title: Effects of Preoperative Oral Carbohydrates Loading in Patients at High Risk of Postoperative Nausea and Vomiting Undergoing Spinal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2015-0984
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Spinal Disease
Keywords: postoperative nausea and vomiting, oral carbohydrate beverage
MeSH Terms: conditions — Spinal Diseases; Postoperative Nausea and Vomiting; Vomiting | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral carbohydrate beverage group (Experimental)
  Interventions: Other: oral carbohydrate beverage
- control group (Placebo Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: oral carbohydrate beverage — oral carbohydrate beverage (12.8% carbohydrates, 50 kcal/100ml, 290 mOsm/kg, NO-NPO®, Daesang WelLife Co., Ltd., Korea) 400ml in the evening of the day before surgery and at 6 am on the day of surgery, respectively
  Arms: oral carbohydrate beverage group
Other: control group — NPO from midnight of the day before surgery
  Arms: control group

SUMMARY:
Many patients receiving opioid based analgesia after spinal surgery experience postoperative nausea and vomiting (PONV) despite prophylaxis and treatment with antiemetic agents. Dehydration caused by fasting prior to surgery is associated with the development of PONV. The aim of this study is to investigate the effect of oral carbohydrates loading prior to surgery in patients at high risk of PONV undergoing spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* female patient between 20 and 65 of age with ASA physical status Ⅰ-Ⅱ
* patient scheduled for elective spine surgery
* no smoking history

Exclusion Criteria:

* hepatorenal disease
* BMI > 35 kg/m2
* gastrointestinal disease
* vomiting within 24h
* administration of antiemetics or opioids within 24 h prior to surgery
* pregnant
* problem with communication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
incidence of nausea and vomiting | 48 hours

SECONDARY OUTCOMES:
severity of nausea | 48 hours
  11-point numerical rating scale (0: no nausea ~10: worst imaginable nausea)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided